CLINICAL TRIAL: NCT05814666
Title: An Open-Label, Phase II, Randomized, Controlled Study of Danvatirsen Plus Pembrolizumab Compared to Pembrolizumab Alone in Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Activity and Safety of Danvatirsen and Pembrolizumab in HNSCC
Acronym: PEMDA-HN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis was negative
Sponsor: Flamingo Therapeutics NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLM-6774-201
Record Dates: First submitted 2023-03-10; First posted 2023-04-18 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — danvatirsen; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Danvatirsen plus pembrolizumab (Experimental): Danvatirsen dosing:
  Week 1: Danvatirsen intravenously (IV) on Days 1, 3, and 5
  Week 2 and subsequent weeks: Danvatirsen IV weekly
  Pembrolizumab dosing:
  Pembrolizumab every 3 weeks after the Danvatirsen dose.
  Interventions: Drug: Danvatirsen; Drug: Pembrolizumab
- Pembrolizumab (Active Comparator): Pembrolizumab IV every 3 weeks
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Danvatirsen — Danvatirsen is a STAT3 targeting drug.
  Other Names: ISIS 481464; AZD9150
  Arms: Danvatirsen plus pembrolizumab
Drug: Pembrolizumab — Pembrolizumab is a monoclonal antibody that binds to the PD-1 receptor and blocks its interaction with PD-L1 and PD-L2
  Other Names: Keytruda

SUMMARY:
Open-label, Phase II, randomized, controlled study evaluating the efficacy and safety of danvatirsen in combination with pembrolizumab compared with pembrolizumab alone as first-line treatment of patients with recurrent/metastatic (R/M) HNSCC. Two-thirds of patients will be randomized to receive danvatirsen and pembrolizumab and one-third will be randomized to receive pembrolizumab alone.

DETAILED DESCRIPTION:
This is a multicenter, open-label, Phase II, randomized, controlled study to determine the efficacy, safety, and other indicators of clinical and biological activity of the combination of danvatirsen and pembrolizumab as first-line treatment for R/M HNSCC.

After providing informed consent, patients will be assessed for eligibility during the screening phase of the study. All patients must be willing and able to provide a formalin fixed paraffin-embedded (FFPE) archival or fresh tumor sample collected during the screening period; a fresh biopsy is preferred if safe and feasible to obtain and consented to by the patient. Following the screening period, eligible patients will be randomized in a 2:1 ratio to danvatirsen + pembrolizumab or pembrolizumab monotherapy, respectively. Patients will receive treatment in 21-day cycles. Patients assigned to the pembrolizumab monotherapy arm will receive treatment until a criterion for discontinuation is met or a maximum of 24 months of treatment. Patients assigned to combination therapy will receive both treatments until a criterion for discontinuation is met or the patient has received a maximum of 24 months of treatment, after which they may remain on danvatirsen monotherapy.

Patients in both treatment arms will have radiologic tumor assessments every 6 weeks (±1 week), regardless of treatment delays, until objective disease progression, initiation of new anticancer treatment, death, withdrawal of consent, or end of study, whichever occurs first.

All patients who discontinue study treatment for any reason will have a safety follow-up visit 30 days (+7 days) after the last dose of study treatment and a follow-up for AEs 90 days (+7 days) after the last dose of pembrolizumab. Patients will be followed for survival at 12 week (±7 days) intervals until death or withdrawal of consent, whichever occurs first. Survival follow-up will continue until at least 15 months after the last patient is randomized in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent (signed and dated).
2. Aged ≥18 years at the time of informed consent.
3. Recurrent/metastatic histologically or cytologically proven squamous cell carcinoma of the head and neck that is considered incurable by local therapy. Eligible primary tumor locations are oropharynx, oral cavity, hypopharynx, and larynx.
4. Presence of measurable tumor per RECIST v1.1 criteria.
5. Detectable PD-L1 expression in tumor, defined as CPS ≥1 determined by a FDA or national regulatory agency of the country in which the patient resides.-approved test.
6. Baseline fresh tumor biopsy or archival specimen.
7. ECOG performance status of 0 or 1.
8. Adequate organ function within 10 days of study treatment,
9. Oxygen saturation on room air ≥92% by pulse oximetry.
10. Females must be non-pregnant and non-lactating and either be postmenopausal or agree to adequate birth control.
11. Males must be surgically sterile or agree to adequate birth control.
12. Has an estimated life expectancy of at least 3 months.
13. Has recovered from all complications or surgery and all toxicities of prior therapy

Exclusion Criteria:

1. Prior therapy for metastatic HNSCC.
2. Has disease suitable for local therapy with curative intent.
3. Primary tumor of the nasopharynx.
4. Has received prior therapy with an anti-programmed death 1 (PD-1), anti PD L1, or anti-programmed death-ligand-2 (PD-L2).
5. Radiation therapy (or other non-systemic therapy) within 2 weeks of Day 1 of study treatment.
6. Known autoimmune disease that has required systemic treatment
7. Known immunodeficiency or receiving systemic steroid therapy that would be the equivalent of >10 mg prednisone daily
8. Prior allogeneic tissue/solid organ transplant.
9. Has significant cardiovascular disease
10. Has received a live vaccine within 30 days
11. Active infection requiring systemic antiviral or antimicrobial therapy
12. History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
13. History of other malignancies
14. Active HIV infection except patients who are currently stable on antiretroviral therapy for at least 4 weeks
15. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
16. Treated or untreated parenchymal brain metastases or leptomeningeal disease.
17. Treatment with another investigational drug, biological agent, or device within 1 month of screening, or 5 half-lives of investigational agent (if known), whichever is longer.
18. Hypersensitivity to any component of danvatirsen or pembrolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Saba, MD, Study Chair — Emory University
Locations (32):
- United States (21):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - University of California Irvine (UCI), Irvine, California
  - TMPN Hunt Cancer Care, Torrance, California
  - University of California Los Angeles, Westwood, Los Angeles, California
  - University of Colorado Hospital (UCH) Anschutz Cancer Pavilion, Aurora, Colorado
  - Miami Cancer Institute, Miami, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - University of Illinois Cancer Center, Chicago, Illinois
  - AMR Kansas City Oncology, Merriam, Kansas
  - University of Kansas Medical Center, Westwood, Kansas
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - University of Maryland Baltimore, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Morristown Medical Center, Morristown, New Jersey
  - Mount Sinai, New York, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - The Christ Hospital Cancer Center, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland, Cleveland, Ohio
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - UT Southwestern Medical Center/Simmons Comprehensive Cancer Center, Dallas, Texas
- South Korea (5):
  - Dong-A University Hospital, Busan
  - Kosin University College of Medicine - Kosin University Gospel Hospital (KUGH), Busan
  - Gyeongsang National University Hospital, Jinju
  - Korea University Medical Center (KUMC), Seoul
  - The Catholic University of Korea - Eunpyeong St. Mary's Hospital, Seoul
- United Kingdom (6):
  - Saint James's University Hospital (SJUH) - St James's Institute of Oncology, Leeds
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Barts Health MHS Trust (Barts and The London NHS Trust) - St Bartholomew's (Barts) Hospital, London
  - The Royal Marsden NHS Foundation Trust, London
  - East and North Hertfordshire NHS Trust, Lister Hospital, Northwood
  - The Royal Marsden NHS Foundation Trust, Sutton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was open from May 2023 through May 2025. Patients were recruited from community based practices, research institutions and universities located in the United States, United Kingdom and South Korea.
  An early assessment of response in patients with CPS ≥1 and <20 was performed and the response rate in this subgroup did not pass the minimum prespecified efficacy level, subsequently eligibility was restricted to patients with CPS ≥20.
Pre-assignment Details: From May 2023 through May 2025, 94 patients were screened, 69 met the eligibility criteria and were randomized. Of the 69 patients that started the treatment period (45 danvatirsen combination arm/24 pembrolizumab arm), 3 patients in the pembrolizumab arm discontinued the study before receiving treatment. 66 patients in total received treatment (45 danvatirsen combination/21 pembrolizumab)
Groups:
- Danvatirsen Plus Pembrolizumab: Danvatirsen dosing:
  Week 1: Danvatirsen intravenously (IV) on Days 1, 3, and 5
  Week 2 and subsequent weeks: Danvatirsen IV weekly
  Pembrolizumab dosing:
  Pembrolizumab every 3 weeks after the Danvatirsen dose.
  Danvatirsen: Danvatirsen is a STAT3 targeting drug.
  Pembrolizumab: Pembrolizumab is a monoclonal antibody that binds to the PD-1 receptor and blocks its interaction with PD-L1 and PD-L2
Period: Overall Study
Arm/Group | Danvatirsen Plus Pembrolizumab | Pembrolizumab
Started (45 pts were randomized to the danva combo arm started and 24 pts were randomized in the pembro arm started however 3 pts in the pembro arm discontinued prior to receiving any doses of pembrolizumab. Therefore the total number of patients that received treatment and included in the safety and efficacy analysis were 45 pt in the danva combo arm and 21 pts in the pembro arm) | 45 | 24
Completed (A total of 48 patients completed treatment per the protocol.) | 34 | 14
Not Completed | 11 | 10
Not completed — Study terminated by Sponsor | 11 | 7
Not completed — Patients withdrew prior to receiving study treatment | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Danvatirsen Plus Pembrolizumab | Pembrolizumab | Total
Number analyzed (Participants) | 45 | 21 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 8 | 27
  >=65 years | 26 | 13 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (11.68) | 65.7 (9.35) | 64.7 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 15
  Male | 34 | 17 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 41 | 19 | 60
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 1 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 24 | 18 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 11 | 0 | 11
  United States | 24 | 18 | 42
  United Kingdom | 10 | 3 | 13
PD-L1 Combined Positive Score (CPS) [Count of Participants; unit: Participants] — All patients were required to have a positive PD-L1 expression determined by a test approved by FDA or the national regulatory agency of the country in which the patient resided to be eligible for enrollment. The PD-L1 measurement was provided as a Combined Positive Score (CPS). The higher the CPS number, the more tumor/immune cells expressing PD-L1. Patients were stratified by their CPS value (<=19 and >=20). The patients with a CPS>= 20 were further categorized.
  Participants
    1-19 | 12 | 7 | 19
    >=20 | 33 | 14 | 47
    20-49 | 12 | 6 | 18
    >=50 | 21 | 8 | 29
Human Papillomavirus (HPV) [Count of Participants; unit: Participants] — HPV status as reported by study sites
  Participants
    Positive | 11 | 5 | 16
    Negative | 20 | 6 | 26
    Unknown | 14 | 10 | 24
Eastern Cooperative Group Performance Status (ECOG [Count of Participants; unit: Participants] — An ECOG Performance Status of 0 (Fully active, able to carry on all pre-disease performance without restriction) or 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature) was required for inclusion in the trial.
  Participants
    ECOG = 0 | 15 | 7 | 22
    ECOG = 1 | 30 | 14 | 44

OUTCOME MEASURES:

1. Primary Outcome: Confirmed ORR
Description: Determine the ORR (Partial response [PR] + CR defined according to RECIST v1.1) as determined by the Investigator for the combination of danvatirsen and pembrolizumab compared with pembrolizumab alone
Time Frame: Up to 18 months
Population: Will include all patients who receive at least 1 dose of study treatment based on the treatment assigned at randomization. 45 pts in the danvatirsen arm were randomized and received at least 1 dose of study treatment, 24 patients in the pembrolizumab arm were randomized however only 21 patients received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Danvatirsen Plus Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 45 | 21
Participants | 7 | 3
Statistical Analysis 1: Comparison: Danvatirsen Plus Pembrolizumab vs Pembrolizumab; Test type: Superiority; p = 0.6039, Fisher Exact — Fisher's Exact 1-Tailed p-value

2. Secondary Outcome: Number of Participants With Adverse Events as Assessed by CTCAE v5.0
Description: Adverse Events are assessed and graded according to Common Toxicity Criteria for Adverse Events (CTCAE) Version 5.0.
Time Frame: Up to 18 months
Population: The Safety Analysis will include all patients who receive at least 1 dose of study treatment based on the actual treatment received. 45 pts in the danvatirsen arm were randomized and received at least 1 dose of study treatment, 24 patients in the pembrolizumab arm were randomized however only 21 patients received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Danvatirsen Plus Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 45 | 21
Participants | 37 | 10

3. Secondary Outcome: DOR
Description: Duration of Response by RECIST v1.1
Time Frame: Up to 18months
Population: Will include all patients who receive at least 1 dose of study treatment and whose best overall response was a CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Danvatirsen Plus Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 7 | 3
Months | 6.36 [5.68 to NA] — There were insufficient events to estimate the specific parameter | NA [NA to NA] — There were insufficient events to estimate the specific parameter

4. Secondary Outcome: DCR & CR Rate
Description: Disease control rate and complete response rate by RECIST v1.1
Time Frame: Up to 18months
Population: Will include all patients that received at least 1 dose of study treatment. 45 pts in the danvatirsen arm were randomized and received at least 1 dose of study treatment, 24 patients in the pembrolizumab arm were randomized however only 21 patients received at least one dose of study treatment. DCR and CR rates will be determined in all patients and within patients with a CPS >=20
Measure: Count of Participants; unit: Participants
Arm/Group | Danvatirsen Plus Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 45 | 21
Participants
  Disease Control Rate (DCR) In all patients | 21 | 12
  Disease Control Rate (DCR) in patients with a CPS>=20: number analyzed (Participants) | 33 | 14
  Disease Control Rate (DCR) in patients with a CPS>=20 | 15 | 9
  Complete Response (CR) Rate in all patients | 1 | 0
  Complete Response (CR) Rate in patients with a CPS>=20: number analyzed (Participants) | 33 | 14
  Complete Response (CR) Rate in patients with a CPS>=20 | 1 | 0

5. Secondary Outcome: ORR in Tumors With CPS ≥20 and ≥ 50
Description: Overall response rate per RECIST v1.1 in tumors with CPS< 20, CPS ≥ 20 and CPS ≥ 50
Time Frame: Up to 18months
Population: Will include all patients who receive at least 1 dose of study treatment based on the treatment assigned at randomization. 45 pts in the danvatirsen arm were randomized and received at least 1 dose of study treatment, 24 patients in the pembrolizumab arm were randomized however only 21 patients received at least one dose of study treatment. ORR will be determined in patients with a CPS< 20, CPS >=20 and CPS>=50.
Measure: Count of Participants; unit: Participants
Arm/Group | Danvatirsen Plus Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 45 | 21
Participants
  In patients with CPS<20: number analyzed (Participants) | 12 | 7
  In patients with CPS<20 | 1 | 0
  In patients with a CPS>=20: number analyzed (Participants) | 33 | 14
  In patients with a CPS>=20 | 6 | 3
  In patients with a CPS>=50: number analyzed (Participants) | 21 | 8
  In patients with a CPS>=50 | 4 | 3

6. Secondary Outcome: DOR in Tumors With CPS ≥20 and ≥50
Description: Duration of response by RECIST v1.1 in tumors with CPS ≥ 20 and ≥50
Time Frame: Up to 18months
Population: Includes only patients that achieved a CR or PR. DOR is defined as the date of the patient's first best overall response of CR or PR to the earliest date of documented progression or to death if no prior evidence of disease progression.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Danvatirsen Plus Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 6 | 3
Months
  In patients with a CPS>=20 | 6.36 [5.68 to NA] — There were insufficient events to estimate the specific parameter. | NA [NA to NA] — There were insufficient events to estimate the specific parameter
  In patients with a CPS>=50: number analyzed (Participants) | 4 | 3
  In patients with a CPS>=50 | 7.03 [NA to NA] — There were insufficient events to estimate the specific parameter. Note that only 4 participants were analyzed, those with a response. Of the 4 responders only 1 had a non-censored value, while the other 3 remained as responders at the time of the analysis cut-off date. With only 1 non-censored value, there is no estimate of variability, and as a result, both confidence interval limits appear as NA. | NA [NA to NA] — There were insufficient events to estimate the specific parameter

7. Secondary Outcome: PFS
Description: Progression-free survival by RECIST v1.1, defined as the time from randomization to the first documentation of progressive disease (PD) or death from any cause, whichever comes first
Time Frame: Up to 18months
Population: PFS will be determined in all patients and in patients with a CPS>=20 who receive at least 1 dose of study treatment.45 pts in the danvatirsen arm were randomized and received at least 1 dose of study treatment, 24 patients in the pembrolizumab arm were randomized however only 21 patients received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Danvatirsen Plus Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 45 | 21
Months
  In all patients | 3.52 [1.48 to 6.83] | 2.92 [1.41 to NA] — There were insufficient events to estimate the specific parameter
  In patients with a CPS>20: number analyzed (Participants) | 33 | 14
  In patients with a CPS>20 | 3.52 [1.35 to 6.83] | NA [NA to NA] — There were insufficient events to estimate the specific parameter

8. Secondary Outcome: OS
Description: Overall survival, defined as time from randomization to death from any cause
Time Frame: Up to 30months
Population: Data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Arm/Group | Danvatirsen Plus Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Maximum Plasma Concentration
Description: Maximum concentration recorded [Cmax]of danvatirsen at defined timepoints in the combination regimen
Time Frame: Up to 18 months
Population: An interim analysis of the Overall Response Rate failed to demonstrate a clinical benefit of danvatirsen. As a result the study was terminated early, all development activities of danvatirsen were discontinued and the PK analysis was not performed. Samples were not analyzed for this pre-specified Outcome Measurement and have since been destroyed therefore no future analysis will occur.
Arm/Group | Danvatirsen Plus Pembrolizumab
Number analyzed (Participants) | 0

10. Secondary Outcome: Trough Concentration
Description: Trough concentration [Ctrough] of danvatirsen at defined timepoints in the combination regimen
Time Frame: Up to 18 months
Population: as for outcome 9
Arm/Group | Danvatirsen Plus Pembrolizumab
Number analyzed (Participants) | 0

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve
Description: Area under the plasma concentration-time curve over the dosing interval [AUCtau] of danvatirsen at defined timepoints in the combination regimen
Time Frame: Up to 18 months
Population: as for outcome 9
Arm/Group | Danvatirsen Plus Pembrolizumab
Number analyzed (Participants) | 0

12. Secondary Outcome: Time to Maximum Plasma Concentration
Description: Time to maximum plasma concentration [Tmax]) after single and multiple doses at defined timepoints in the combination regimen
Time Frame: Up to 18 months
Population: as for outcome 9
Arm/Group | Danvatirsen Plus Pembrolizumab
Number analyzed (Participants) | 0

13. Secondary Outcome: Immunogenicity of Danvatirsen
Description: Anti-danvatirsen antibody titers at defined timepoints in the combination regimen
Time Frame: Up to 18 months
Population: An interim analysis of the Overall Response Rate failed to demonstrate a clinical benefit of danvatirsen. As a result the study was terminated early, all development activities of danvatirsen were discontinued and the ADA analysis was not performed. Samples were not analyzed for this pre-specified Outcome Measurement and have since been destroyed therefore no future analysis will occur.
Arm/Group | Danvatirsen Plus Pembrolizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Approximately 25 months
Description: AEs from first dose through 30 days after the last dose and 90 days after the last dose of pembrolizumab or until the patient began a new anticancer treatment were reported in the CRF. All AEs and SAEs that occur from the signing of the ICF until the first dose of study treatment were recorded in the CRF only if the event was related to a study procedure.
Groups:
- Pembrolizumab: Pembrolizumab IV every 3 weeks after the Danvatirsen dose.
  Pembrolizumab: Pembrolizumab is a monoclonal antibody that binds to the PD-1 receptor and blocks its interaction with PD-L1 and PD-L2
Arm/Group | Danvatirsen Plus Pembrolizumab | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 8/45 | 4/21
Serious Adverse Events (participants affected / at risk) | 25/45 | 6/21
Other Adverse Events (participants affected / at risk) | 44/45 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Danvatirsen Plus Pembrolizumab (N=45) | Pembrolizumab (N=21)
Leukaemoid reaction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 3 (3) | 2 (2)
Death (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Swelling face (General disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 1 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrong product administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Vasogenic cerebral oedema (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Danvatirsen Plus Pembrolizumab (N=45) | Pembrolizumab (N=21)
Anaemia (Blood and lymphatic system disorders) | 14 (40) | 4 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (12) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (11) | 0 (0)
Hypothyroidism (Endocrine disorders) | 5 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 9 (12) | 4 (4)
Nausea (Gastrointestinal disorders) | 10 (12) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (10) | 2 (2)
Vomiting (Gastrointestinal disorders) | 7 (10) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 5 (6) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 0 (0)
Fatigue (General disorders) | 17 (25) | 8 (10)
Pyrexia (General disorders) | 3 (4) | 0 (0)
Secretion discharge (General disorders) | 3 (3) | 1 (1)
Asthenia (General disorders) | 3 (3) | 0 (0)
Chills (General disorders) | 1 (1) | 2 (2)
Disease Progression (General disorders) | 3 (3) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 6 (10) | 0 (0)
Pneumonia (Infections and infestations) | 6 (8) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (4) | 0 (0)
Pneumonia Aspiration (Infections and infestations) | 4 (6) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 19 (50) | 0 (0)
Platelet count decreased (Investigations) | 8 (32) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 16 (30) | 0 (0)
Weight decreased (Investigations) | 3 (11) | 3 (3)
White blood cell count decreased (Investigations) | 6 (10) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (7) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (11) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (4)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 1 (1)
Dizziness (Nervous system disorders) | 3 (4) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (2)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data is owned by the Sponsor. Sponsor shall have right to first publication of the results of the Study. PI may publish after 18 months of study termination if no publication by the sponsor. Sponsor may have up to 120 days to review the publication and has the right for confidential information to be removed.

DOCUMENTS (2):
  • Study Protocol (2025-05-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT05814666/Prot_000.pdf
  • Statistical Analysis Plan (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT05814666/SAP_001.pdf